CLINICAL TRIAL: NCT02837120
Title: Retrospective Study of Acute Chest Pain in Extremely Critical Condition for More Than Ten Years
Acronym: RESPECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 201671respect
Record Dates: First submitted 2016-07-07; First posted 2016-07-19 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myocardial Infarction; Pulmonary Embolism; Aortic Dissection
Keywords: retrospective study; acute myocardial infarction; acute aortic dissection; pulmonary embolism; unstable angina
MeSH Terms: conditions — Pulmonary Embolism; Aortic Dissection; Angina, Unstable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Acute non-traumatic chest pain is a common kind of symptom in extremely critical condition, with various pathogenesis and different level of risk . Chest pain in high risk takes 1/3 of that. It mainly includes acute coronary syndrome (including myocardial infarction and unstable angina pectoris, accounted for over 95% of chest pain in high risk), aortic dissection, pulmonary embolism etc, and is in high lethality and deformity.

The investigators do the research :

1. To study the diagnosis and management condition of acute chest pain in extremely critical condition for last ten or more years in Qilu Hospital,Shandong University.
2. To discuss the significance of key accompanying symptoms(for example radiating pain, chest distress, sweating, nausea etc), physical signs and lab examination in early diagnosis and risk stratification of acute chest pain in extremely critical condition.
3. To study the effect factors of thrombus burden in STEMI patients, at the same time, creat a a simple, practical and scientific method of blood clots classification.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of Qilu Hospital, whose electronic medical records were searched out by terms of acute myocardial infarction, aortic dissection, pulmonary embolism and unstable angina in International Classification of Diseases(ICD)-10 code from Jan.2003 to Sep.2015.

Exclusion Criteria:

* Patients whose medical records are false, omitted or uncompleted because of transference, death et al.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in Qilu Hospital with high risk chest pain diseases(acute myocardial infarction, aortic dissection, pulmonary embolism, unstable angina) from 2003.01 to 2015.09
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and management of acute chest pain diseases in extremely critical condition | A week after data collected
  In-hospital mortality, hospitalization days

SECONDARY OUTCOMES:
Clinical characteristics of participants for demographics, medical history, examination results and investigations retrieved from electronic medical records | A week after data collected
  Frequency of chest pain, sweating, nausea, radiating pain, dyspnea and temperature, pulse, respiration rates, blood pressure, value of blood glucose, D-Dimer, et al, on admission.
The predicted factors of thrombus burden in STEMI patients, and the influence of thrombus burden on mortality | A week after data collected
  The relationship between value of leukocyte,glucose,lipid,blood pressure et al, all-cause mortality and thrombus burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China